CLINICAL TRIAL: NCT04192825
Title: Analysis of Therapeutic Management Strategies for Anal Suppurations of Crohn's Disease
Acronym: 3T-LAP
Status: Recruiting | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC18_8808_3T-LAP
Record Dates: First submitted 2019-12-05; First posted 2019-12-10 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Crohn Disease; Anal Suppurations; Drainage Procedure
MeSH Terms: conditions — Crohn Disease | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: surgical treatment — surgical drainage and/or surgical reconstruction procedures to anoperineal suppurations according to the doctor's decision

SUMMARY:
Determine the optimal therapeutic combination associated with complete clinical and anatomical remission of anal suppurations of Crohn's disease at 12 months.

DETAILED DESCRIPTION:
The management of anoperineal suppurations of Crohn's disease is most often based on clinical practice recommendations, the results of randomized controlled trials and also the analysis of monocentric cohort studies from expert centres. In these latter studies, there is an overall improvement in patients during follow-up with a high level of satisfaction (two thirds of cases), often assessed by the operator himself or the clinician who provides therapeutic management. The most striking finding is the one that highlights the use of combined therapeutic strategies combining immunosuppressants, biotherapies, antibiotics, surgical drainage and surgical reconstruction procedures to varying degrees. Thus, the absence of fistula pathway flow in the long term is the consequence of both maintenance treatment with biotherapies and several surgical procedures. When the characteristics of fistula pathways considered healed on clinical examination are analysed by MRI exploration, an active unhealed pathway persists in two thirds of cases, again emphasizing the inadequacy of clinical examination as a means of assessing recovery. For this reason, fistula pathway closure strategies do not provide much greater benefit than simple removal of the drainage loop. Conversely, medical treatment optimization strategies based on MRI evaluation of the therapeutic response have demonstrated high efficacy. It is necessary to (re)define the therapeutic management of patients with anoperineal lesions. This strategy must be based on a better initial stratification of patients based on prognostic factors derived from available scientific data. A second step consists in setting therapeutic efficacy objectives that take into account the control of the inflammatory component of anal Crohn's disease and the preservation of the anatomical and functional capital of the anus. Only a large prospective cohort at the national level provides the opportunity to study these prognostic factors and to specify the level of optimal therapeutic responses

ELIGIBILITY:
Inclusion Criteria:

* Persons over 18 years of age
* People suffering from anal suppuration of Crohn's disease for whom a drainage procedure is planned.
* Person who has received written and oral information about the protocol and has not expressed opposition to participate in the study.

Exclusion Criteria:

* No one who is unable to have an anesthetic, structural or psychological examination by MRI and/or surgery.
* Person planning a planned absence that could hinder participation in the research (travel abroad, relocation, impending transfer);
* Person with an associated pathology that is a priority for care;
* Vulnerable person (minors, persons under guardianship or curatorship, or deprived of their liberty by a judicial or administrative decision

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Person suffering from anal suppuration related to Crohn's Disease
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2025-08-03 (Estimated); Study Completion 2028-08-03 (Estimated)

PRIMARY OUTCOMES:
Clinical and anatomical healing | 12 months.
  The healing of anal fistula is defined by the combination of two criteria at 12 months :
  * MRI criteria = absence of a T2 hyper signal from the path(s) AND the absence of an abscess AND
  * Complete clinical response = no pain, no discharge, and no drain

CONTACTS AND LOCATIONS:
Overall Officials: Laurent SIPROUDHIS, PH-PD, Principal Investigator — Rennes University Hospital
Locations (1):
- Centre Hospitalier de Rennes, Rennes, France